CLINICAL TRIAL: NCT02201394
Title: Normalizing Platelet Reactivity After Treatment With Ticagrelor
Brief Title: Reversing Ticagrelor's Effects With Fresh Platelets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Juan J Badimon, Director, AtheroThrombosis Research Unit; Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1802
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: Antiplatelet; Ticagrelor; Platelets; Thrombosis; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loading dose (Experimental): Patients with stable CVD given a single ticagrelor loading dose and aspirin loading dose
  Interventions: Drug: Ticagrelor loading dose; Drug: Aspirin loading dose
- Maintenance dose (Experimental): Patients with stable CVD given ticagrelor maintenance dose and aspirin maintenance dose for one week.
  Interventions: Drug: Ticagrelor maintenance dose; Drug: Aspirin maintenance dose

INTERVENTIONS:
Drug: Ticagrelor loading dose — Single loading dose of Ticagrelor 180 mg
  Other Names: Brilinta
  Arms: Loading dose
Drug: Aspirin loading dose — Single loading dose of Aspirin 325 mg
  Other Names: Acetylsalicylic acid; ASA
  Arms: Loading dose
Drug: Ticagrelor maintenance dose — Ticagrelor 90 mg twice daily x 7 days
  Other Names: Ticagrelor; Brilinta
  Arms: Maintenance dose
Drug: Aspirin maintenance dose — Aspirin 81 mg once daily x 7 days
  Other Names: Aspirin; ASA
  Arms: Maintenance dose

SUMMARY:
Acute coronary syndrome (ACS) patients treated with antiplatelet drugs who require coronary artery bypass grafting (CABG) surgery have to wait 5-7 days for the effects of the drugs to wean off. This treatment-devoid period leaves the patient vulnerable, therefore any means to shorten this period could be useful. The present study aims to investigate the possibility of reversing the antiplatelet effects of ticagrelor with the help of fresh donor platelets. Fresh platelets will be added to blood samples of treated patients in varying concentrations at specific timepoints to determine the time and amount of fresh platelets needed to normalize platelet reactivity in the treated samples.

DETAILED DESCRIPTION:
The current American College of Cardiology/American Heart Association (ACC/AHA) guidelines for ACS patients requiring CABG surgery after treatment with dual antiplatelet therapy recommend delaying surgery for 5-7 days after discontinuation of therapy, to allow for the dissipation of its antiplatelet effects. This treatment-devoid waiting period puts the ACS patients at risk for further cardiovascular events. Any means to shorten this vulnerable period would be of critical value. One possibility to speed up the recovery of the inhibited platelets is to administer infusions of fresh platelets. In fact, platelet transfusions are frequently administered to patients during surgery who had received prior antiplatelet therapy. However, the degree to which these transfusions restore platelet function in the recipient subjects' blood and the time from dosing when they are most effective are unknown. The timing is critical in scenarios where urgent surgery is required because infusion of platelets too soon after antiplatelet dosing could render them useless by the residual drug in circulation.

The aim of the present study is to investigate the restoration of platelet function of ticagrelor-treated subjects by adding donor platelets to their blood. The study would have 2 arms mimicking different clinical scenarios:

1. Clinical Scenario 1 - Patient given a loading dose (LD) of ticagrelor in the emergency room, requires surgery: A single LD of ticagrelor (180 mg) with aspirin (325 mg) will be given to study subjects and platelet testing will be performed after addition of fresh platelets to their blood ex vivo. Donor platelets will be added at 4-, 6-, 24- and 48-hours post-dose, to assess the time required for normalizing subject's platelet function after a LD of ticagrelor.
2. Clinical Scenario 2 - Patient on maintenance dosing (MD) of ticagrelor, requires surgery: Subjects will receive ticagrelor (90 mg twice daily) with aspirin (81 mg once daily) for 3-7 days. After the last dose, platelet testing will be performed after addition of fresh platelets to their blood ex vivo, at 4-, 6-, 24- and 48-hours post-dose to assess the time required for normalizing subject's platelet function after daily treatment with ticagrelor.

Platelet testing will be carried out using the following methodologies:

1. Platelet Aggregation - VerifyNow P2Y12 assay.
2. Platelet Aggregation - Multiplate Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteer between 18 and 75 years old.
* History of stable (i.e. non-acute) cardiovascular disease or the presence of risk factors for cardiovascular disease (i.e. hypertension, diabetes, hyperlipidemia, high calcium score and abnormal findings on angiography or stress test).

Exclusion Criteria:

* Conditions associated with hemorrhagic risk, e.g., frequent epistaxis, gastrointestinal ulcer, hemorrhagic vascular lesions, recent surgery.
* Allergy or hypersensitivity to aspirin or ticagrelor.
* Loss of >400 mL blood or blood donation within past 3 months.
* Positive serology for hepatitis B (HBs Ag) or hepatitis C.
* History of drug abuse or alcohol abuse.
* Positive pregnancy test.
* Evidence of unstable or acute cardiovascular disease (e.g., unstable angina, recent myocardial infarction, congestive heart failure).
* History of clinically relevant pulmonary, hepatic, gastrointestinal, renal, metabolic, hematologic, neurologic, respiratory or psychiatric disease, bleeding, acute infectious disease or signs of acute illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Badimon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Zafar MU, Smith DA, Baber U, Sartori S, Chen K, Lam DW, Linares-Koloffon CA, Rey-Mendoza J, Jimenez Britez G, Escolar G, Fuster V, Badimon JJ. Impact of Timing on the Functional Recovery Achieved With Platelet Supplementation After Treatment With Ticagrelor. Circ Cardiovasc Interv. 2017 Aug;10(8):e005120. doi: 10.1161/CIRCINTERVENTIONS.117.005120. PMID 28768756

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Stable CVD: DAPT loading dose (Ticagrelor (180 mg) + ASA (325 mg)); DAPT maintenance therapy (Ticagrelor (90 mg BID) + ASA (81 mg OD), for one week (in same patients)
Period: Loading Dose
Arm/Group | Patients With Stable CVD
Started | 20
Completed | 20
Not Completed | 0
Period: Maintenance Dose
Arm/Group | Patients With Stable CVD
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Stable CVD
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Diabetic [Count of Participants; unit: Participants] | 15
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 30.7 (4.5)
Hypertension [Count of Participants; unit: Participants] | 16
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 127.2 (17.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 70.6 (9.0)
Hypercholesterolemia [Count of Participants; unit: Participants] | 19
Cholesterol level [Mean (Standard Deviation); unit: mg/dL] | 158.7 (62.0)
Triglycerides level [Mean (Standard Deviation); unit: mg/dL] | 165.4 (91.4)
LDL level [Mean (Standard Deviation); unit: mg/dL] — low-density lipoprotein
  mg/dL | 85.6 (51.7)
HDL [Mean (Standard Deviation); unit: mg/dL] — high-density lipoprotein
  mg/dL | 42.5 (12.6)
Smoking History [Count of Participants; unit: Participants]
  Current | 2
  Past | 8
  Never | 10
Alcohol Use [Count of Participants; unit: Participants]
  Current | 9
  Past | 3
  Never | 8

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Unit (PRU)
Description: Platelet function normalization using different concentrations (0%, 25%, 50%, and 75% supplementations) of fresh platelet within 48 hours of Ticagrelor Loading dose/last Maintenance dose, assessed using VerifyNow and expressed as P2Y12 Reaction Unit (PRU). The P2Y12 reaction unit (PRU) is an arbitrary unit of measure that represents the amount of platelet aggregation specific to the P2Y12 receptor.
Time Frame: Baseline (pre-treatment), 4, 6, 24 and 48 hours post Loading dose/last Maintenance dose
Population: Patients with stable CVD
Measure: Mean (Standard Deviation); unit: PRU
Groups:
- Loading Dose: Ticagrelor (180 mg) + ASA (325 mg).
- Maintenance Dose: Ticagrelor (90 mg BID) + ASA (81 mg OD), for one week
Arm/Group | Loading Dose | Maintenance Dose
Number analyzed (Participants) | 20 | 20
PRU
  Baseline | 284.1 (42.2) | 284.1 (42.2)
  Post-dose 4 hours 0% | 39.1 (25.9) | 37.5 (32.4)
  4 hours 25% | 69.6 (35.6) | 72.2 (38.5)
  4 hours 50% | 100.3 (49.6) | 88.4 (42.9)
  4 hours 75% | 98.6 (54.4) | 85.9 (49.4)
  Post-dose 6 hours 0% | 25.9 (28.9) | 24.0 (30.3)
  6 hours 25% | 55.3 (50.2) | 46.0 (37.3)
  6 hours 50% | 67.8 (53.8) | 55.4 (41.8)
  6 hours 75% | 71.2 (42.8) | 67.7 (45.3)
  Post-dose 24 hours 0% | 127.6 (58.8) | 119.0 (78.0)
  24 hours 25% | 157.3 (52.5) | 147.6 (65.2)
  24 hours 50% | 165.9 (40.5) | 158.0 (43.5)
  24 hours 75% | 162.5 (29.4) | 154.0 (51.0)
  Post-dose 48 hours 0% | 250.6 (45.8) | 214.8 (74.0)
  48 hours 25% | 249.5 (35.1) | 219.7 (52.2)
  48 hours 50% | 226.2 (51.6) | 221.2 (44.2)
  48 hours 75% | 204.2 (45.9) | 203.9 (41.5)

2. Primary Outcome: Platelet Aggregation Using Multiplate Analyzer
Description: Platelet function normalization using different concentrations of fresh platelet within 48 hours of Ticagrelor Loading dose/last Maintenance dose, assessed using Multiplate Aggregometry (ADPtest), results expressed as Area Under Curve (U), where 1 U = 10 AU * min.
Time Frame: Baseline (pre-treatment), 4, 6, 24, and 48 hours post Loading dose/last Maintenance dose
Population: Patients with stable CVD
Measure: Mean (Standard Deviation); unit: 10 AU * min
Arm/Group | Loading Dose | Maintenance Dose
Number analyzed (Participants) | 20 | 20
10 AU * min
  Baseline (pre-dose | 67.0 (14.3) | 67.0 (14.3)
  Post-dose 4 hours 0% | 13.6 (4.6) | 15.7 (6.7)
  4 hours 25% | 18.7 (5.2) | 20.9 (6.1)
  4 hours 50% | 21.4 (7.7) | 22.1 (5.9)
  4 hours 75% | 23.6 (8.4) | 24.2 (6.3)
  Post-dose 6 hours 0% | 12.3 (5.9) | 13.4 (6.0)
  6 hours 25% | 17.3 (6.1) | 16.5 (5.5)
  6 hours 50% | 20.7 (6.5) | 18.9 (6.3)
  6 hours 75% | 22.3 (7.5) | 20.4 (6.2)
  Post dose 24 hours 0% | 24.9 (14.0) | 25.6 (15.6)
  24 hours 25% | 39.7 (18.1) | 35.5 (15.1)
  24 hours 50% | 49.3 (17.9) | 43.3 (16.7)
  24 hours 75% | 52.8 (22.7) | 47.5 (18.2)
  Post-dose 48 hours 0% | 41.3 (17.7) | 39.1 (21.3)
  48 hours 25% | 57.7 (17.6) | 56.8 (19.5)
  48 hours 50% | 68.6 (20.4) | 63.8 (19.1)
  48 hours 75% | 72.8 (18.4) | 70.3 (23.0)

ADVERSE EVENTS:
Arm/Group | Patients With Stable CVD
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Study design is partly in vitro as testing of study aims (reversing effects of antiplatelet therapy by adding fresh platelets in different concentrations and at different times) would be nearly impossible using an in vivo study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes